CLINICAL TRIAL: NCT05473260
Title: Home Monitoring Vs. Hospitalization for Mild Acute Pancreatitis. A Pilot Randomized Controlled Clinical Trial
Brief Title: Home Monitoring Vs. Hospitalization for Mild Acute Pancreatitis
Acronym: RHINO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, BUSQUETS, JULI, Digestive and General Surgeon, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RHINO-TRIAL
Record Dates: First submitted 2022-07-11; First posted 2022-07-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Acute Pancreatitis
Keywords: acute pancreatitis; mild pancreatitis; outpatient protocol
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOSPI Group (Active Comparator): Patients with mild acute pancreatitis randomized to in-hospital care.
  Interventions: Other: Control
- HOME Group (Experimental): Patients with mild acute pancreatitis randomized to early discharge and outpatient clinic follow-up.
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Control — In-patient care.
  Other Names: HOSPIT
  Arms: HOSPI Group
Other: Experimental — Early discharge and outpatient follow-up.
  Other Names: HOME
  Arms: HOME Group

SUMMARY:
Acute pancreatitis accounts for a large number of hospital admissions every year. Some studies have shown that early oral feeding protocols are safe, and one previous study suggests the possibility of home care for mild acute pancreatitis.

DETAILED DESCRIPTION:
Approximately 80% of all cases of acute pancreatitis are mild and only require supportive care for pain and nausea control and an adequate fluid replacement. Currently, all patients in our setting diagnosed with mild acute pancreatitis are admitted to a conventional hospitalization ward under the supervision of the Digestive and General Surgery Department or the Gastroenterology Department. Symptomatic treatment is administered, and abdominal ultrasound is performed to assess the cause of pancreatic inflammation. The remaining 20% fulfill the severity criteria from its onset onwards and require intensive care support.

We will conduct a multicenter randomized controlled clinical trial to compare two different approaches to mild non-alcoholic acute pancreatitis: hospital admission and outpatient management.

ELIGIBILITY:
INCLUSION CRITERIA

Patients diagnosed with mild acute pancreatitis based on at least two of the three following criteria:

* Abdominal pain
* Amylase or lipase 3x ULN (in blood/urine)
* Imaging tests (Ultrasound/CT scan) suggestive of acute pancreatitis.

Age ≥18 years and <80 years

Absence of potential pancreatitis-related severity criteria:

* No evidence of SIRS in the emergency room
* C-Reactive Protein levels <150mg/dL
* Marked increase in the White Blood Cell Count
* Absence of coagulopathy (INR <1.4)
* Hematocrit < 44%
* Creatinine < 170 µmol/L
* BISAP score ≤2 at the time of randomization.

Patients with good pain response to 12-hour supportive care in the ER (VAS <4) or adequate oral feeding tolerability.

Absence of local or systemic complications of acute pancreatitis on imaging tests.

Adequate cognitive capacity and without any previous diagnose of psychiatric disease.

Patients who meet each participating hospital home care criteria. Patients who give their written informed consent to participate.

EXCLUSION CRITERIA

Past medical history of pancreatic disease:

* Known or newly diagnosed chronic pancreatitis (Wirsung dilation or pancreatic calcifications in previous imaging tests)
* Patients with recurrent acute pancreatitis (>3 episodes/year) or an episode of acute pancreatitis <1 month ago.
* Acute pancreatitis after endoscopic retrograde cholangiography.
* Hyperbilirubinemia >3x ULN

Comorbidities that required previous hospitalization (myocardial infarction, liver cirrhosis, chronic kidney disease, or chronic lung disease).

BMI ≥35 Kg/m2 Patients who refuse to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2025-07-16 (Estimated); Study Completion 2025-07-16 (Estimated)

PRIMARY OUTCOMES:
7-day (after randomization) treatment failure rate | 7 days
  Treatment failure is defined as a VAS >3 and/or oral feeding intolerance (nausea, repeated vomiting episodes, early satiety).

SECONDARY OUTCOMES:
Cumulative incidence of complications secondary to acute pancreatitis during the first 30 days after diagnosis | 30 days
  Complications include, but are not limited to, abscess formation, pseudocysts, local necrosis, kidney failure, respiratory failure.
Hospital readmission during the first 30 days after diagnosis | 30 days
  Number of patients readmitted to the hospital during the first 30 days after diagnosis.
Cumulative incidence of mortality during the first 30 days after diagnosis | 30 days
  30-day mortality
Estimated costs of each intervention | 7 days
Median (95%CI) Charlson Comorbidity Score per group | 7 days
Median (95%CI) EuroQoL 5 Dimensions Quality of Life Score | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided